CLINICAL TRIAL: NCT03528252
Title: Effectiveness of Written Dietary Advice on Lipoproteins - a Pragmatic Randomized Controlled Trial (MYDICLIN)
Brief Title: Effectiveness of Written Dietary Advice on Lipoproteins - a Pragmatic Randomized Controlled Trial
Acronym: MYDICLIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Dalarna County Council, Sweden (Other)
Responsible Party: Principal Investigator, David Iggman, General practitioner, Principal Investigator, Associated researcher, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MYDICLIN; Dnr 2018/119 (Other: Uppsala Regional Ethics Committee)
Record Dates: First submitted 2018-04-19; First posted 2018-05-17 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Cholesterol, LDL
Keywords: cholesterol; LDL cholesterol; Triglycerides; Diet; Food; Lipoproteins
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Two identical parallel groups
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization by sealed envelopes, opened in private. Allocation sequence and envelopes provided by external agent. Participants are instructed not to discuss intervention outside household. No more than one (randomly selected) participant per household allowed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LDL Cholesterol (Active Comparator): Will receive dietary advice effective for reducing LDL cholesterol.
  Interventions: Other: Written advice LDL Cholesterol
- Triglycerides (Sham Comparator): Will not be aware that they are in fact Control Group. Will receive dietary advice effective for reducing Triglycerides, but neutral for LDL cholesterol.
  Interventions: Other: Written advice Triglycerides

INTERVENTIONS:
Other: Written advice LDL Cholesterol — One A4 paper with written information on both sides
  Other Names: Active Intervention
  Arms: LDL Cholesterol
Other: Written advice Triglycerides — One A4 paper with written information on both sides
  Other Names: Control Group
  Arms: Triglycerides

SUMMARY:
This study investigates the effect of detailed, written dietary advice for improving blood lipids, in a primary care setting. n=222 participants will be randomized to Active Intervention or Control Group. After 3 weeks' intervention, participants will receive written feedback on the effect on their blood lipids. After 6 months, another blood sample is drawn and participants will receive further written feedback.

DETAILED DESCRIPTION:
The Active Intervention Group will receive detailed dietary advice based on current evidence for food choices that improve LDL cholesterol levels. The information will contain motivational strategies, e.g. "It's great that you want to improve your blood lipids! What are your three main reasons that you want to improve your blood lipids? What food choices suit you? How low can you go?" Participants will receive a table of ten suggested healthy food choices and be instructed to mark for each day a certain food change has been made.

The Control Group will receive similar advice and motivational strategies, with the one difference being the dietary advice, that will focus on Triglycerides instead of LDL cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Listed patient at Svärdsjö Primary Health Care Centre
* Willing to reduce blood lipids

Exclusion Criteria:

* Drugs affecting blood lipids (statins, ezetimibe, fibrates, PCSK9-inhibitors, neuroleptic drugs, cortisone, amiodarone, estrogen, progesterone, testosterone, cyclosporin, tacrolimus, loop diuretics, protease inhibitors and anti-convulsants; whereas beta blockers, thiazide diuretics, and SGLT2-inhibitors are allowed under established medication
* Current malignant disease
* Extreme diet
* Abnormal metabolism e.g. uncontrolled hypothyroidism
* Dementia
* Unability to comprehend written information in Swedish
* Other participant from same household
* Current employment on Svärdsjö Primary Health Care Centre

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
LDL Cholesterol | 3 weeks and 6 months
  Change in plasma LDL Cholesterol levels

SECONDARY OUTCOMES:
Total Cholesterol | 3 weeks and 6 months
  Change in plasma Total Cholesterol levels
HDL Cholesterol | 3 weeks and 6 months
  Change in plasma HDL Cholesterol levels
Apolipoproteins | 3 weeks and 6 months
  Change in plasma Apolipoprotein levels
Success rate | 3 weeks and 6 months
  Percentage of participants that reduce LDL Cholesterol at least 10%
Responder effect | 6 months and 3 weeks, respectively
  Change in plasma LDL cholesterol after 6 months in participants that reduce LDL Cholesterol at least 10% at 3 weeks
Double sampling requirement | 3 weeks and 6 months
  Number of participants that would have been misclassified if not double sampling hade been performed for LDL cholesterol
Cost of intervention | 3 weeks and 6 months
  Cost of intervention, in comparison to possible health gains
Effective food choices | 3 weeks and 6 months
  Food choices that are in practice effective for lowering LDL cholesterol
Stated reasons | 3 weeks and 6 months
  Stated reasons for wanting to improve blood lipid profile and associations with effect on LDL Cholesterol
PSCK9 | 3 weeks and 6 months
  Change in serum PCSK9 levels
Lipoprotein(a) | 3 weeks and 6 months
  Change in plasma lipoprotein(a) levels

CONTACTS AND LOCATIONS:
Overall Officials: David Iggman, M.D. Ph.D, Principal Investigator — Uppsala University
Locations (1):
- Svärdsjö Primary Health Care Centre, Falun, Dalarna County, Sweden

IPD SHARING:
Plan to Share IPD: No
N/A, data sharing is not included in Ethics application. Further consent from participants may be required.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT03528252/SAP_000.pdf
  • Study Protocol (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT03528252/Prot_001.pdf